CLINICAL TRIAL: NCT04227782
Title: MRI and Stable Isotope Tracer Studies for Detecting the Progression of Non-Alcoholic Steatohepatitis (NASH)
Acronym: MRI-Detect
Status: Active, not recruiting | Type: Observational
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Other Study IDs: MRI-DETECT
Record Dates: First submitted 2019-12-19; First posted 2020-01-14 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2023-11

CONDITIONS: Non-Alcoholic Fatty Liver Disease
Keywords: magnetic resonance spectroscopy; magnetic resonance imaging; isotope tracer studies; fatty acid oxidation; de-novo lipogenesis; liver phosphorus MR spectroscopy
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Magnetic Resonance Imaging; Positron-Emission Tomography

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum, plasma, urine
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- NAFLD
  Interventions: Diagnostic Test: Magnetic Resonance Imaging; Other: Stable Isotope Study
- NASH
  Interventions: Diagnostic Test: Magnetic Resonance Imaging; Other: Stable Isotope Study
- Cirrhosis
  Interventions: Diagnostic Test: Magnetic Resonance Imaging; Other: Stable Isotope Study
- Healthy Volunteers
  Interventions: Diagnostic Test: Magnetic Resonance Imaging

INTERVENTIONS:
Diagnostic Test: Magnetic Resonance Imaging — Magnetic Resonance Imaging
  Other Names: magnetic resonance spectroscopy
Other: Stable Isotope Study — Stable Isotope study
  Groups: Cirrhosis; NAFLD; NASH

SUMMARY:
One-third of the world's population suffers from Non-Alcoholic Fatty Liver Disease (NAFLD), that is a disease with an accumulation of fat in the liver. Some patients with NAFLD will progress in their disease to develop inflammation, scarring of the liver tissue, and cirrhosis that can lead to liver failure. The mechanisms of the disease and its progression are still not fully understood. It is therefore critical to find early markers that can identify the patients that will progress so that they can be treated early.

A compound called L-carnitine, synthesised in the body from two amino acids; lysine and methionine, is critical for fat metabolism. Some studies have shown that it is decreased in liver disease patients and that L-carnitine supplementation can protect the liver function.

This study aims to increase the understanding of the mechanisms behind NAFLD disease progression through its different stages. This may help diagnostic methods to be developed to predict the patients at risk for developing severe liver disease. Furthermore, fat metabolism and L-carnitine levels will be established in the different disease stages to evaluate whether fat metabolism could be compromised.

Magnetic Resonance Imaging (MRI) will be used for imaging of the whole liver and the heart to investigate metabolism and function non-invasively. Whole-body metabolism and how carbohydrates are taken up from diets are converted to fats in the body will be explored using stable isotope labelling. This study will recruit 30 participants with NAFLD; 10 each for low-risk NALFD, biopsy-proven NASH and compensated NASH cirrhosis. Participants will undergo MRI, followed by a stable isotope labelled study, where through blood- and breathe samples, metabolism will be investigated.

An additional 10 healthy participants will be assessed using MR techniques to assess whether an injection of L-carnitine can lead to increase of L-carnitine in the liver such that it can be detected by MR. This is to validate a methodology prior to using it in NAFLD participants.

DETAILED DESCRIPTION:
STUDY 1: Functional and Metabolic Parameters in participants with NAFLD Participants will undertake two study visits, within a 14-day period. One of the visits will involve MR assessments that will take up to three hours in total. The second visit will involve a postprandial study day using stable isotopes. Baseline samples will be taken from participants, and after they have been fed a standardised test meal to assess whole-body and liver specific postprandial metabolism - this visit will last up to eight hours.

Magnetic Resonance Imaging (MRI) and Spectroscopy (MRS) and stable isotope labelling are two methodologies to investigate in vivo metabolism and function non-invasively. MRI gives information about liver structure and tissue composition, and heart function. MRS can also evaluate tissue energetics and composition using spectroscopy. Stable isotope-labelling studies allow for the measurement of whole-body fatty acid oxidation and de-novo lipogenesis in the pre- and post-prandial state. These two methodologies will be used in our study to evaluate participants with different severity of NAFLD and could help elucidate how the disease progresses.

STUDY 2: MRI evaluation of L-carnitine In parallel to study 1, the physiological response to L-carnitine (50 mg/kg i.v.) will be investigated only in healthy participants with 1H MRS.

These participants will only take part in one visit, during which they will undergo a baseline MRI scan, followed by the injection of L-carnitine. The MRI/MRS will be repeated two hours after the injection. AC has previously been measured in skeletal muscle using 1H MRS. In this study it will be measured in the septum of the heart and in the liver pre and 2 hours post-injection of 50 mg/kg i.v. of L-carnitine.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18
* In cases where histologic evidence is needed, the pathologist evaluation of a liver biopsy should be obtained within 90 days prior to screening.

Participants with simple steatosis

* Liver biopsy that shows features of simple steatosis and no signs of advanced fibrosis or NASH (F3) or cirrhosis (F4). Simple steatosis will be defined as the presence of lipid inclusions in ≥ 5% of hepatocytes without both of lobular inflammation and hepatocyte ballooning. Steatosis with either lobular inflammation or ballooning will be included in this category provided there is no bridging fibrosis (<F3 on the NASH CRN fibrosis classification system), OR
* Findings of fatty liver on ultrasound in patients with low risk of NASH or advanced fibrosis defined as liver stiffness measurement <8kPa.

Participants with NASH:

o Liver biopsy that shows presence of all the features of NASH (≥ 5% steatosis, lobular inflammation and hepatocyte ballooning) and without liver cirrhosis. Low-grade fibrosis are allowed.

Participants with NASH cirrhosis:

* Liver biopsy that shows features of NASH cirrhosis. Historical liver biopsies will be acceptable provided there has been no significant weight loss (> 5% of body weight) between the time of biopsy and recruitment, OR
* Presence of metabolic comorbidities and clinical (stigmata of chronic liver disease), radiological (e.g. irregular liver edge, features of portal hypertension), laboratory (deranged clotting, low platelet count) and non-invasive test results consistent with liver cirrhosis (e.g. liver stiffness >20kPa).

Exclusion Criteria:

* The participant may not enter the study if ANY of the following apply:

For the albumin1 infusion: At screening individuals are asked about any allergies and in excluded to the albumin infusion in case of egg allergy. In case of lactose intolerance, milk will be exchanged to a lactosefree non-dairy form.

* Contraindication to MRI
* History of alcoholism or a greater than recommended weekly alcohol intake (14 units per week)
* Liver disease other than NAFLD (chronic viral hepatitis B or C, autoimmune liver disease, primary biliary cholangitis, primary sclerosing cholangitis, haemochromatosis, Wilson's disease, alpha 1 antitrypsin deficiency, drug induced liver injury)
* Pregnant/Planning to get pregnant
* Low haemoglobin (NAFLD participants), women with Hb < 11g/l and men with Hb <12g/l will be excluded
* Unwillingness to refrain from blood donations in the specified period (NAFLD participants)
* Extensive tattooing covering the MRI scanning area

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Population is patients with Non-alcoholic Fatty Liver Disease (NAFLD), either with simple steatosis, NASH or cirrhosis
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Differences in whole-body fatty acid oxidation in a stable isotope labelled postprandial study day in participant groups. | baseline
  Changes in the incorporation of 13C (from dietary fat or sugar) into CO2 measured using a breath analyser, as a marker of whole-body dietary fatty acid/glucose oxidations.To explore whole-body fatty acid oxidation in individuals with simple steatosis, NASH and NASH with Cirrhosis

SECONDARY OUTCOMES:
Intrahepatic fatty acid synthesis in a stable isotope labelled postprandial study day in participant groups | baseline
  Differences in hepatic fatty acid synthesis as measured by incorporation of 2H2 palmitate from 2H2O into very low density lipoprotein triglyceride (VLDL-TG) in participants with simple steatosis, NASH and NASH Cirrhosis.
Cardiac Function using MRI in participant groups | baseline
  Comparison of the cardiac function as assessed by ejection fraction
Difference in liver metabolites using MRS in participant groups | baseline
  Differences in hepatic energetics using 31P MRS comparing Pi/ATP ratio in participants with simple steatosis, NASH and NASH Cirrhosis.
Difference in heart metabolites using MRS in participant groups | baseline
  Differences in cardiac fat content using 1H MRS in participants with simple steatosis, NASH and NASH Cirrhosis.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Oxford, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Savic D, Mozes FE, Green PG, Burrage MK, Kjaer MS, Hodson L, Neubauer S, Pavlides M, Valkovic L. Detection and alterations of acetylcarnitine (AC) in human liver by 1 H MRS at 3T after supplementation with l-carnitine. Magn Reson Med. 2023 Apr;89(4):1314-1322. doi: 10.1002/mrm.29544. Epub 2022 Dec 27. PMID 36573435